CLINICAL TRIAL: NCT06508840
Title: Clear Conversations: Evaluating a Verbal Health Literacy Intervention in Derbyshire
Brief Title: The Clear Conversations Project
Status: Recruiting | Type: Observational
Sponsor: University of Sheffield (Other)
Collaborators: Derbyshire Community Health Services NHS Foundation Trust (Unknown); Debyshire County Council (Unknown)
Responsible Party: Sponsor
Other Study IDs: 185136; 336469 (Other: IRAS)
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-07

CONDITIONS: COPD; Weight Loss
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Rehab Programme: Pulmonary Rehab Programme staff and patients. The five physiotherapists who deliver the programmes will receive Verbal Health Literacy training and implementation support.
  Patients will enrol and complete the Pulmonary Rehab programme as usual. That is two sessions a week for six weeks.
  Interventions: Other: Verbal Health Literacy training session
- Weight Management Programme: Six out of twelve Health Improvement Advisors, who deliver the programmes, will receive Verbal Health Literacy Training and implementation support.
  Service users will attend the programme as usual. That is one session a week for 12 weeks.
  Interventions: Other: Verbal Health Literacy training session

INTERVENTIONS:
Other: Verbal Health Literacy training session — Five respiratory physiotherapists and half (6/12) weight management programme advisors, will receive a two hour Verbal Health Literacy training session. The training session will focus on three techniques: simple language, 'Teachback' and 'Chunk and check'. They will also receive implementation support from a Health Literacy Officer.
  All pulmonary rehab patients will attend programmes run by physiotherapists trained in Verbal Health Literacy techniques.
  Weight management programme service users will attend programmes run by trained and untrained staff.

SUMMARY:
Understanding health information can be difficult. This means some people struggle to know how to manage their health. Also, people may not know what health services to use or when to use them. This can lead to poorer health.

It is therefore important health workers can communicate information clearly. This is so people using health services can understand it and know what to do. Having clear conversations with service users could help them to improve their health. More research is needed into this area. This is so we can understand and improve health conversations.

In this research project health workers will be provided with training. The training will teach them ways to improve their communication skills. Health workers will also receive support from a Health Literacy Officer. The Investigators want to see if this can improve service user outcomes and reduce health inequalities.

The investigators will ask health workers and service users from a Local Authority and an NHS service to take part. Service users will attend the health programmes as normal. Staff who have and have not received the training will deliver the programmes.

The investigators will ask service users to complete questionnaires. The investigators will also collect service user data from the programmes. This data will be collected before and after they attend. The investigators will compare this data with the previous year.

The investigators will observe health workers delivering the programmes. The investigators will use a check list to see how they use the skills they have learnt. The investigators will ask health workers to complete a questionnaire before and after they attend the training. The investigators will run focus groups with the health workers six months later. The investigators want to understand if the training was useful. The investigators also want to know if the health workers are using the skills they learnt in their practice.

DETAILED DESCRIPTION:
Health Literacy is important so people can understand how to access healthcare services and receive and understand the help that they need.

It is known that people who struggle to understand health information often have lower education levels and are from poorer areas. They are likely to have worse health outcomes.

Interventions to improve Health Literacy should be aimed at those with lower levels of education, living in poorer parts of the country or with a long term health condition or disability.

In Derbyshire six out of ten people and three out of nine areas are thought to be below the UK average for reading and maths. It is therefore important to address Health Literacy in this region to improve the health of the region and reduce health inequalities.

Research to improve people's Health Literacy has been undertaken. Most of these studies have focused on written health information. Studies that have focused on Verbal (communication) Health Literacy skills have only looked at short term outcomes. They have also failed to focus on how healthcare staff can use the skills in practice.

This research will aim to understand if the investigators can improve healthcare staff's verbal communication skills. This is so service users can understand advice and instructions they are given. So, they feel able to act on the advice and instructions to improve their health. Healthcare staff will receive training on Verbal (communication) Health Literacy techniques. They will receive support from a Health Literacy Officer. This is to help them use the techniques they learn in the training in their practice.

A number of different outcomes will be measured to answer the studies objectives. These will focus on understanding:

1. Staffs perceptions of the training;
2. Staff's knowledge, skills and confidence to use the techniques in their practice;
3. Service users subjective Health Literacy and activation skills
4. Service and service user outcomes

This will be a mixed methods evaluation. It will include a process evaluation to understand the acceptability and feasibility of the training session. Pre and post test and controlled pre and post test evaluation of health outcomes will also be measured.

The research will be undertaken in two different services:

1. A local authority run Weight Management Programme. This service is led by eight Health Improvement Advisors. They deliver the advice and education sessions. The sessions run face to face and online over a 12 week rolling period. Service users attend one session a week for 12 weeks.
2. A NHS Pulmonary Rehabilitation Programme. The service is led by six physiotherapists and two specialist nurses. They deliver the exercise, advice and education sessions. The sessions take place face to face for 6 weeks. Service users attend two sessions a week for six weeks. It is also a rolling programme.

Half of the Health Improvement Advisors from the Weight Management Programme will receive the two hour Verbal Health Literacy training. This means a controlled pre and post test evaluation will be undertaken with this service.

Six physiotherapists who deliver the Pulmonary Rehabilitation Programme will receive the two hour Verbal Health Literacy training. A pre and post test evaluation only will be undertaken for this service.

Follow on support from a Health Literacy Officer will be offered to all trained staff. This is to help them use the skills they have learnt in their practice.

Service users who enrol onto the two programmes during the research period will be invited to take part.

A summary participant information sheet will be made available in the first instance. This will either be given to all those who enrol by the member of staff in charge of enrolment. Or it will be included, along with an electronic consent form via a link in the the services enrolment/welcome email. Full project information sheets will be made available to all those wanting to find out more.

The following data will be collected from staff in order to answer the projects objectives.

1. Pre and post intervention staff questionnaires. These will be completed at baseline, immediately after attending the training and then 8 weeks later. All staff that attend Verbal Health Literacy training during the period of the research will be asked to complete the questionnaires. That is not just staff from the two participating services. Their purpose is to understand:

   * Staffs levels of Verbal Health Literacy knowledge before the training;
   * How useful staff found the training;
   * How confident staff feel to use the techniques in their practice;
   * Any additional support staff participants may require to help them use the techniques in their practice.

   The training and questionnaires are part of routine staff professional development. The questionnaires are distributed via a NHS microsoft teams form by the Health Literacy Officer who delivers the training. They will be distributed in the same way during the research period.
2. Pre and post intervention observations or session recordings. A checklist will be completed. This is to see how staff are using the Verbal Health Literacy techniques in their practice.

   Half of the weight management service, who will receive the training, and the six physiotherapists from the pulmonary rehabilitation service will be observed or their sessions recorded. One session for each recruited member of staff will be observed or recorded and a checklist completed by the lead researcher before they attend the training. Where audio recording is the preferred or most practical method an encrypted audio-recorder will be used.

   One session for each recruited member of staff will be observed or recorded 12-16 weeks after they have received the training and a checklist completed. This is to see if staff are still using the techniques in their practice.
3. Focus group interviews. Focus group interviews will be carried out with all of the trained staff from the two services where possible. Two focus groups, one for weight management service staff and one for pulmonary rehabilitation staff, will take place 4-6 months after staff have attended the training. The focus groups will supplement the questionnaire data. They will provide deeper and richer insights into staff thoughts and perceptions about the training itself and how they have been able to use the techniques (or not) in their practice.

The focus groups will take place during staff training time. They will take place either face to face or via videocall. Face to face focus groups will be audio recorded, using an encrypted audio recorded.

Videocalls will take place via googlemeet. They will be recorded and transcribed via the googlemeet recording and transcribing functions. All recordings and or transcriptions will be downloaded to secure University of Sheffield file stores. Original recordings will deleted from the audio recorder immediately and from the google drive after google transcripts have been checked.

Audio recorded recordings will be transcribed using University of Sheffield approved transcribers. All transcripts will be pseudonymised. This is so they are private and participants can not be identified.

Consent will be gained from all staff prior to completing:

* The questionnaires,
* Being observed or recorded,
* Attending a focus group interview. Individual service user and aggregate service and health outcome data will also be collected. This is so the investigators can see if training staff improves service and health outcomes.

Service users who enrol on the two programmes during the period of the research will be asked to:

1. Complete a Health Literacy Questionnaire.

   They will be asked to complete this:
   * when they enrol on the programme,
   * when they have completed the programme. That is at 12 weeks for weight management, and at 6 weeks for pulmonary rehabilitation.

   Consent will be gained from all service users prior to completing the questionnaire.

   The Health Literacy Questionnaires will be distributed in one of two ways. Either by email invitation via an electronic link. This will direct participants to the Qualtrics version of the questionnaire.

   Qualtrics is an online survey platform approved by the University of Sheffield Information Governance.

   Or they will be sent to participants in the post. The completed postal questionnaires will be returned to the researcher via a stamped addressed envelope.
2. Service users will be asked to consent to share their data that is routinely collected by the programme they attend.

   The primary outcomes that will be measured and collected will be:
   * Weight in Kg for the weight management programme
   * The Chronic Respiratory Disease Questionnaire (CRDQ) for the pulmonary rehabilitation programme.

   The secondary outcomes will be:
   * The short form Warwick and Edinburgh Mental Health and Wellbeing Scale (weight management).
   * the timed shuttle walking test (in meters), the LINK Questionnaire, GAD-7, PHQ-9, strength test (pulmonary rehabilitation).

   Individual demographic data will also be collected. Such as, age, gender, ethnicity and postcode.
3. Grouped data from both services will be collected, such as:

   * Summarised demographic data eg. age, gender, ethnicity, IMD.
   * Programme attendance rates.
   * Average weight loss.
   * Average changes CRDQ. We aim to reach a sample size of approximately 252 service users for the weight management programme. That is approximately 126 whose programme is delivered by trained staff and approximately 126 whose programme is delivered by non trained staff.

We aim to achieve a sample of 72 service users for the pulmonary rehabilitation. This will be achieved by collecting data from two, six week cohorts of the programme. These calculations are based on minimum and maximum potential attendees and likely consent/return rates.

This summarised data will be collected during the three month period of the research. For example, May-July 2024. It will also be collected from a similar period in 2023.

We estimate that a sample size of 252 will be required for this grouped data for the weight management programme.

This is based upon an estimated mean weight loss of 4.09kg. In order to achieve statistical power to detect small differences in the pulmonary rehabilitation population we are likely to have to extend this request for data to a six month rather than three month period.

We are likely to need to collect data over a 6 month period , that is four, six week cohorts, for the pulmonary rehabilitation programme in order to achieve statistical power.

A patient and public and healthcare professional partnership groups have helped in the design and development of the study documents including:

* The project summary.
* Consent forms.
* Project information sheets. They will continue to be involved to help guide the different stages of the study

ELIGIBILITY:
Inclusion Criteria:

* • Public Health Intervention Advisors delivering the tier 2 weight management programme across Derbyshire.

  * Physiotherapists and specialist nurses involved in the assessment of patients and delivery of the six week DCHS NHS pulmonary rehabilitation programme.
  * Adults aged 18 or over who start the rolling 12 week tier two weight management programme during the intervention period.
  * Adults aged 18 or over, with Chronic Obstructive Pulmonary Disease, who are being assessed for and undertaking the six week pulmonary rehabilitation programme during the study intervention period.
  * For the staff questionnaire only - Healthcare staff from other services that attend Verbal Health Literacy training, during the study period in 2024, will also be eligible

Exclusion Criteria:

* • Service users attending the two service programmes outside of the data collection period.

  * Other pulmonary rehabilitation staff. i.e. staff who are not physiotherapists or specialist nurses.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Physiotherapists and Health Improvement Advisors working in the pulmonary rehab programme and weight management programme respectively.
  Patients/services users attending either of the two programmes during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Chronic Respiratory Disease Questionnaire (CDRQ) | 0, 6 weeks
  The CRQ is an interviewer-administered questionnaire measuring both physical and emotional aspects of chronic respiratory disease. The total score for the CRDQ ranges from 0 to 100, with higher scores indicating better HRQOL
Weight in kilogrammes | 0, 12, 26 weeks
  Services attending the weight management programme will be weighed at the start and end of the programme

SECONDARY OUTCOMES:
The short Warwick and Edinburgh Mental Health and Well being Scale (weight management programme only) | 0 and 12 weeks
  A 7 point scale to enable the monitoring of mental wellbeing in the general population and the evaluation of projects, programmes and policies which aim to improve mental wellbeing. The total score range for SWEMWBS is 7-35. A higher score indicating better HRQL.
Incremental shuttle walking test in meters (Pulmonary Rehab prgramme only) | 0, 6 weeks
  The patient is required to walk around two cones set 9 metres apart (so the final track is 10 metres) in time to a set of auditory beeps. The patient walks for as long as they can until they are either too breathless or can no longer keep up with the beeps, at which time the test ends.
Lung Information Needs Questionnaire (LINQ) - pulmonary rehab programme | 0, 6 weeks
  A brief questionnaire completed prior to the clinical encounter would assist health professionals identify areas of information need. The total score range is 0-25.A higher score indicates a greater need for information.
Generalised Anxiety Disorder Assessment (GAD-7) - Pulmonary rehab programme | 0, 6 weeks
  A self-administered patient questionnaire used as a screening tool and severity measure for generalised anxiety disorder. It measures severity of anxiety, mainly in outpatients.. The total score range is 0-21. A higher score indicating higher levels of anxiety.
Patient Health Questionnaire (PHQ-9) - Pumonary rehab programme | 0-6weeks
  a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders.1 The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care. The total score range is 0-27. A higher score indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Grindell, PhD, Principal Investigator — University of Sheffield
Locations (2):
- United Kingdom (2):
  - Derbyshire County Council, Matlock, Chesterfield
  - Derbyshire Community Health Services NHSFT, Chesterfield, Derbyshire

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of anonymised data on request from the PI

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT06508840/Prot_SAP_000.pdf